CLINICAL TRIAL: NCT01330511
Title: Simplified Diagnostic Algorithm for Evaluation of Neonates With Prenatally Detected Hydronephrosis
Status: Completed | Type: Observational
Sponsor: Rush University Medical Center (Other)
Responsible Party: Farahnak Assadi, MD, RUSH University Medical Center, Pediatrics, Department of Nephrology
Other Study IDs: 10020402
Record Dates: First submitted 2011-04-01; First posted 2011-04-07 (Estimated); Last update posted 2011-04-07 (Estimated); Status verified 2011-04

CONDITIONS: Congenital Hydronephrosis
Keywords: Newborn infant; Congenital hydronephrosis; Postnatal imaging evaluation; Diagnostic algorithm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Bilateral Hydronephrosis Grade I-II: Patients with Bilateral Hydronephrosis Grade I-II
- Bil. Hydronephrosis Grade III-IV, Other: Patient with Bilateral Hydronephrosis Grade III-IV and others with any hydronephrosis and distended bladder or MCKD
- Unilateral Hydronephrosis Grade I-II: Patients with Unilateral Hydronephrosis Grades I-II
- Unilateral Hydronephrosis Grade III-IV: Patients with Unilateral Hydronephrosis Grade III-IV

SUMMARY:
Patients with congenital hydronephrosis will be identified by inpatient consultations performed by Dr. Assadi for congenital hydronephrosis and by outpatient problem lists with congenital hydronephrosis of Dr. Assadi's existing patients. Given standard evaluation will be evaluated to determine if based on initial ultrasound classification an algorithm can be developed to target evaluation studies for the initial evaluation. With a goal of targeting the few children that have need of additional intervention and minimizing the studies performed on children who will spontaneously resolve.

DETAILED DESCRIPTION:
Patients with congenital hydronephrosis will be identified by inpatient consultations performed by Dr. Assadi for congenital hydronephrosis and by outpatient problem lists with congenital hydronephrosis of Dr. Assadi's existing patients. Once identified, the patient's grade of hydronephrosis will be recorded from initial ultrasound based on Society of Fetal Urology (SFU) classification. If no initial SFU classification was assigned to the hydronephrosis a pediatric radiologist will review the initial ultrasound images and classify the grade of hydronephrosis based upon SFU criteria. The patients ensuing evaluation of their hydronephrosis that took place will then be recorded and de-identified. Data to be collected will include: Ultrasound evaluations of the abdomen, retroperitoneum, or renal system, Voiding Cysto-Urethrogram (VCUGs), nuclear studies: diuretic enhanced technetium-99m dietylene triamine penta-acetic acid renogram (DTPA) or technetium-99m Mercapto-acetyl-triglycine renogram (MAG3), referral to pediatric urology for pyeloplasty, serum electrolytes, Blood Urea Nitrogen (BUN) and creatinine, urinalysis, urinary tract infections, and placement on long-term antibiotic prophylaxis.

The follow up evaluation that took place for each patient will then be compared to our proposed algorithm for congenital hydronephrosis evaluation and treatment. This algorithm will be designed based on clinical experience of expert opinion and literature review of each step in the evaluation and treatment. Primary outcomes will be progressive renal function decline and progression to referral to a pediatric urologist for pyeloplasty. Secondary outcomes will be incidence of urinary tract infections and placement on long term antibiotic prophylaxis for urinary tract infection prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for the study were confirmation of the diagnosis of prenatal hydronephrosis by postnatal renal ultrasound

Exclusion Criteria:

* prior history of UTI
* diagnosis of cystic renal dysplasia with poorly functioning kidney
* previous operation on the urinary tract system
* and other deformities of the external genital organs or anomalies in cardiopulmonary and central nervous system

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants with prenatally diagnosed hydronephrosis by ultrasound who have consulted pediatric nephrology
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2005-01; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
surgical intervention required | Follow for minimum 1 year, approximately 2 years goal
  Primary outcome will be progressive renal function decline and progression to referral to a pediatric urologist for pyeloplasty.

CONTACTS AND LOCATIONS:
Overall Officials: Farahnak Assadi, MD, Principal Investigator — RUSH University, Pediatrics, Nephrology
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Background] Warady BA, Chadha V. Chronic kidney disease in children: the global perspective. Pediatr Nephrol. 2007 Dec;22(12):1999-2009. doi: 10.1007/s00467-006-0410-1. Epub 2007 Feb 20. PMID 17310363
- [Background] Mong Hiep TT, Ismaili K, Collart F, Van Damme-Lombaerts R, Godefroid N, Ghuysen MS, Van Hoeck K, Raes A, Janssen F, Robert A. Clinical characteristics and outcomes of children with stage 3-5 chronic kidney disease. Pediatr Nephrol. 2010 May;25(5):935-40. doi: 10.1007/s00467-009-1424-2. Epub 2010 Feb 11. PMID 20148340
- [Background] Ardissino G, Dacco V, Testa S, Bonaudo R, Claris-Appiani A, Taioli E, Marra G, Edefonti A, Sereni F; ItalKid Project. Epidemiology of chronic renal failure in children: data from the ItalKid project. Pediatrics. 2003 Apr;111(4 Pt 1):e382-7. doi: 10.1542/peds.111.4.e382. PMID 12671156
- [Background] Smith JM, Stablein DM, Munoz R, Hebert D, McDonald RA. Contributions of the Transplant Registry: The 2006 Annual Report of the North American Pediatric Renal Trials and Collaborative Studies (NAPRTCS). Pediatr Transplant. 2007 Jun;11(4):366-73. doi: 10.1111/j.1399-3046.2007.00704.x. PMID 17493215
- [Background] Brown T, Mandell J, Lebowitz RL. Neonatal hydronephrosis in the era of sonography. AJR Am J Roentgenol. 1987 May;148(5):959-63. doi: 10.2214/ajr.148.5.959. PMID 3034009
- [Background] Palmer LS, Maizels M, Cartwright PC, Fernbach SK, Conway JJ. Surgery versus observation for managing obstructive grade 3 to 4 unilateral hydronephrosis: a report from the Society for Fetal Urology. J Urol. 1998 Jan;159(1):222-8. doi: 10.1016/s0022-5347(01)64072-2. PMID 9400485
- [Background] Grignon A, Filion R, Filiatrault D, Robitaille P, Homsy Y, Boutin H, Leblond R. Urinary tract dilatation in utero: classification and clinical applications. Radiology. 1986 Sep;160(3):645-7. doi: 10.1148/radiology.160.3.3526402.
- [Background] Anderson N, Clautice-Engle T, Allan R, Abbott G, Wells JE. Detection of obstructive uropathy in the fetus: predictive value of sonographic measurements of renal pelvic diameter at various gestational ages. AJR Am J Roentgenol. 1995 Mar;164(3):719-23. doi: 10.2214/ajr.164.3.7863901.
- [Background] Maizels M, Reisman ME, Flom LS, Nelson J, Fernbach S, Firlit CF, Conway JJ. Grading nephroureteral dilatation detected in the first year of life: correlation with obstruction. J Urol. 1992 Aug;148(2 Pt 2):609-14; discussion 615-6. doi: 10.1016/s0022-5347(17)36668-5. PMID 1640535
- [Background] Fernbach SK, Maizels M, Conway JJ. Ultrasound grading of hydronephrosis: introduction to the system used by the Society for Fetal Urology. Pediatr Radiol. 1993;23(6):478-80. doi: 10.1007/BF02012459. PMID 8255658
- [Background] Conway JJ, Maizels M. The "well tempered" diuretic renogram: a standard method to examine the asymptomatic neonate with hydronephrosis or hydroureteronephrosis. A report from combined meetings of The Society for Fetal Urology and members of The Pediatric Nuclear Medicine Council--The Society of Nuclear Medicine. J Nucl Med. 1992 Nov;33(11):2047-51. PMID 1432172
- [Background] Herndon CD, McKenna PH, Kolon TF, Gonzales ET, Baker LA, Docimo SG. A multicenter outcomes analysis of patients with neonatal reflux presenting with prenatal hydronephrosis. J Urol. 1999 Sep;162(3 Pt 2):1203-8. doi: 10.1016/S0022-5347(01)68134-5. PMID 10458467
- [Background] Ismaili K, Avni FE, Piepsz A, Wissing KM, Cochat P, Aubert D, Hall M. Current management of infants with fetal renal pelvis dilation: a survey by French-speaking pediatric nephrologists and urologists. Pediatr Nephrol. 2004 Sep;19(9):966-71. doi: 10.1007/s00467-004-1506-0. Epub 2004 Jul 6. PMID 15241673
- [Background] Lee JH, Choi HS, Kim JK, Won HS, Kim KS, Moon DH, Cho KS, Park YS. Nonrefluxing neonatal hydronephrosis and the risk of urinary tract infection. J Urol. 2008 Apr;179(4):1524-8. doi: 10.1016/j.juro.2007.11.090. Epub 2008 Mar 4. PMID 18295269
- [Background] Keays MA, Guerra LA, Mihill J, Raju G, Al-Asheeri N, Geier P, Gaboury I, Matzinger M, Pike J, Leonard MP. Reliability assessment of Society for Fetal Urology ultrasound grading system for hydronephrosis. J Urol. 2008 Oct;180(4 Suppl):1680-2; discussion1682-3. doi: 10.1016/j.juro.2008.03.107. Epub 2008 Aug 16. PMID 18708207
- [Background] Yerkes EB, Adams MC, Pope JC 4th, Brock JW 3rd. Does every patient with prenatal hydronephrosis need voiding cystourethrography? J Urol. 1999 Sep;162(3 Pt 2):1218-20. doi: 10.1016/S0022-5347(01)68138-2. PMID 10458470
- [Background] Wiener JS, O'Hara SM. Optimal timing of initial postnatal ultrasonography in newborns with prenatal hydronephrosis. J Urol. 2002 Oct;168(4 Pt 2):1826-9; discussion 1829. doi: 10.1097/01.ju.0000030859.88692.dd. PMID 12352369
- [Background] Docimo SG. Re: Optimal timing of initial postnatal ultrasonography in newborns with prenatal hydronephrosis. J Urol. 2003 Apr;169(4):1474; author reply 1474. doi: 10.1097/01.ju.0000053374.59414.58. No abstract available. PMID 12629390
- [Background] Yang Y, Hou Y, Niu ZB, Wang CL. Long-term follow-up and management of prenatally detected, isolated hydronephrosis. J Pediatr Surg. 2010 Aug;45(8):1701-6. doi: 10.1016/j.jpedsurg.2010.03.030. PMID 20713223
- [Background] Sidhu G, Beyene J, Rosenblum ND. Outcome of isolated antenatal hydronephrosis: a systematic review and meta-analysis. Pediatr Nephrol. 2006 Feb;21(2):218-24. doi: 10.1007/s00467-005-2100-9. Epub 2005 Dec 17. PMID 16362721
- [Background] Estrada CR, Peters CA, Retik AB, Nguyen HT. Vesicoureteral reflux and urinary tract infection in children with a history of prenatal hydronephrosis--should voiding cystourethrography be performed in cases of postnatally persistent grade II hydronephrosis? J Urol. 2009 Feb;181(2):801-6; discussion 806-7. doi: 10.1016/j.juro.2008.10.057. Epub 2008 Dec 17. PMID 19095265
- [Background] Moorthy I, Joshi N, Cook JV, Warren M. Antenatal hydronephrosis: negative predictive value of normal postnatal ultrasound--a 5-year study. Clin Radiol. 2003 Dec;58(12):964-70. doi: 10.1016/s0009-9260(03)00171-5. PMID 14654029
- [Background] Maizels M, Alpert SA, Houston JT, Sabbagha RE, Parilla BV, MacGregor SN. Fetal bladder sagittal length: a simple monitor to assess normal and enlarged fetal bladder size, and forecast clinical outcome. J Urol. 2004 Nov;172(5 Pt 1):1995-9. doi: 10.1097/01.ju.0000142136.17222.07. PMID 15540775
- [Background] Homsy YL, Saad F, Laberge I, Williot P, Pison C. Transitional hydronephrosis of the newborn and infant. J Urol. 1990 Aug;144(2 Pt 2):579-83; discussion 593-4. doi: 10.1016/s0022-5347(17)39527-7. PMID 2197440
- [Background] Peters CA, Skoog SJ, Arant BS Jr, Copp HL, Elder JS, Hudson RG, Khoury AE, Lorenzo AJ, Pohl HG, Shapiro E, Snodgrass WT, Diaz M. Summary of the AUA Guideline on Management of Primary Vesicoureteral Reflux in Children. J Urol. 2010 Sep;184(3):1134-44. doi: 10.1016/j.juro.2010.05.065. Epub 2010 Jul 21. PMID 20650499